CLINICAL TRIAL: NCT05750251
Title: Effect of Upper Eyelid Surgeries on Corneal Topography, Corneal High-order Aberration, Corneal Biomechanical Properties, and Corneal Epithelial Thickness
Brief Title: Effect of Upper Eyelid Surgeries on Corneal Characteristics
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202211048RINA
Record Dates: First submitted 2023-02-06; First posted 2023-03-01 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2023-02

CONDITIONS: Eyelid Diseases; Ptosis, Eyelid
Keywords: Blepharoplasty
MeSH Terms: conditions — Eyelid Diseases; Blepharoptosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ptosis patient: Undergo conventional ptosis correction surgery, including levator muscle resection surgery and Müller's muscle-conjuctival resection surgery
  Interventions: Procedure: levator muscle resection surgery; Procedure: Müller's muscle-conjuctival resection surgery
- Eyelid retraction patient: Undergo conventional ptosis correction surgery, including full-thickness anterior blepharotomy surgery
  Interventions: Procedure: full-thickness anterior blepharotomy surgery

INTERVENTIONS:
Procedure: levator muscle resection surgery — conventional ptosis surgery
  Groups: Ptosis patient
Procedure: Müller's muscle-conjuctival resection surgery — conventional ptosis surgery
  Groups: Ptosis patient
Procedure: full-thickness anterior blepharotomy surgery — conventional eyelid retraction surgery
  Groups: Eyelid retraction patient

SUMMARY:
The goal of this prospective observational study is to learn about the impact of conventional eyelid correction surgery on the eye's health and function in ptosis and eyelid retraction patient. The main questions it aims to answer are: •

1. Changes in corneal topography, higher-order corneal aberrations, corneal biomechanical characteristics, and corneal epithelial thickness before and after the surgery
2. Influence of corneal refraction examinations , vision change, and tear film function after the surgery

Fifty participants will undergo conventional eyelid correction surgery by the same ophthalmologist (YH Wei) and non-invasive examinations before and after the surgery. The patient will be separate to 2 groups, including 30 with correction for ptosis and 20 with correction for eyelid retraction. The research will collect information of the operated eye and fellow eye, and the data will be compared between operated and fellow eye and with the other group.

DETAILED DESCRIPTION:
The position of the upper eyelid affects the health and function of the eye. Ptosis can obstruct the vision, and eyelid retraction can result in the loss of proper protection of the ocular surface. Through conventional upper eyelid correction surgery, the height of the upper eyelid can be adjusted to a proper position. However, after upper eyelid surgery, the pressure of the upper eyelid on the corneal surface may change, affecting corneal topography, higher-order corneal aberrations, corneal biomechanical characteristics, and corneal epithelial thickness. These changes may affect postoperative vision and visual quality. The impact of upper eyelid surgery on corneal refraction and corneal biomechanical characteristics remains inconclusive in current studies, and the impact on corneal epithelial thickness is even less investigated. This is a prospective observational study, expecting to enroll 50 patients who have undergone upper eyelid surgery, including 30 for ptosis correction and 20 for eyelid retraction correction. Non-invasive examinations will be used to assess changes in corneal topography, higher-order corneal aberrations, corneal biomechanical characteristics, and corneal epithelial thickness before and after the surgery to understand the impact of upper eyelid surgery on the ocular surface and the possible mechanism or influencing factors of postoperative vision changes.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* marginal reflex distance 1 (MRD1) ≦ 2-2.5 mm
* levator muscle function (LMF) ≧ 8 mm

Group 2:

* with upper scleral show

Exclusion Criteria:

* pregnancy
* previous corneal surgery
* with corneal scar
* pterygium
* keratoconus
* significant ocular surface disease
* wearing rigid contact lens

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from 20-year-old to 80-year old who need eyelid correction surgery, Group 1 : Ptosis patient with marginal reflex distance 1 (MRD1) ≦ 2-2.5 mm and levator muscle fundction (LMF) ≧ 8 mm; Group 2 : Eyelid retraction patient with upper scleral show. The population excluded patients with pregnancy, previous corneal surgery, corneal scar, pterygium, keratoconus, significant ocular surface disease, or wearing rigid contact lens.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Change from best corrected visual acuity at 3 months after the surgery | Baseline, Month 1, Month 3
  Assess best corrected visual acuity by qualified optometrists, with Landolt C chart-based examination Record as decimal visual acuity
Change from intraocular pressure at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure intraocular pressure with tonometers in unit of mmHg
Change from eyeball axial length at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure eyeball axial length with A-scan in unit of mm
Change from slit lamp examination at 3 months after the surgery | Baseline, Month 1, Month 3
  Assess local findings with a slit lamp by same and only ophthalmologist, Dr. YH Wei
Change from margin to reflex distance (MRD) at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure margin to reflex distance with a ruler in unit of mm by same and only ophthalmologist, Dr. YH Wei MRD-1: from the corneal light reflex to the level of the center of the upper-eyelid margin MRD-2: from the corneal light reflex to the central portion of the lower eyelid
Change from levator muscle function (LMF) at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure levator muscle function with a ruler in unit of mm by same and only ophthalmologist, Dr. YH Wei LMF: the distance the eyelid travel from downgaze to upgaze while the frontalis muscle is held inactive at the brow
Change from lagophthalmos at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure lagophthalmos with a ruler in unit of mm by same and only ophthalmologist, Dr. YH Wei
Change from basal tear volume at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure basal tear volume with Schirmer's test in unit of mm/5 minutes Schirmer's test: small paper strip with rulers printed is placed over the temporal one-third of the lower lid margin and inserted inside the inferior conjunctival fornices under local infiltrating anesthesia. The strips are removed after 5 minutes and the amount of tears produced in that time is measured by reading off of the length of wetting in millimeters.
Change from ocular surface disease index (OSDI) at 3 months after the surgery | Baseline, Month 1, Month 3
  Interview participants with OSDI questionnaire to assesses dry eye symptoms and the effects on vision-related function by same and only ophthalmologist, Dr. YH Wei
Change from tear break up time at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure tear break up time with Oculus Keratograph 5M (OCULUS, Wetzlar, Germany) in unit of sec
Change from corneal biomechanical characteristics at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure corneal biomechanical characteristics with Oculus Corvis ST tonometer (OCULUS, Wetzlar, Germany)
Change from corneal topography at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure corneal topography with Tomey TMS topographer (TOMEY, Nuremberg, Germany) and record as topography map.
Change from higher-order corneal aberrations at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure higher-order corneal aberrations with Tracey iTrace wavefront aberrometer and corneal topography (TRACEY, Texas, USA), using beam of light projected into the eyes. The wavefront of the reflected light is captured by the machine and collected the distortion and aberration of the cornea.
Change from corneal epithelial thickness at 3 months after the surgery | Baseline, Month 1, Month 3
  Measure corneal epithelial thickness with anterior segment optical coherence tomography in unit of micrometer (Visionix USA, Illinois, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsuan Wei, PhD, Study Chair — National Taiwan University Hospital, Department of Ophthalmology
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Aksu Ceylan N, Yeniad B. Effects of Upper Eyelid Surgery on the Ocular Surface and Corneal Topography. Turk J Ophthalmol. 2022 Feb 23;52(1):50-56. doi: 10.4274/tjo.galenos.2021.63255. PMID 35196840
- [Background] Savino G, Battendieri R, Riso M, Traina S, Poscia A, D'Amico G, Caporossi A. Corneal Topographic Changes After Eyelid Ptosis Surgery. Cornea. 2016 Apr;35(4):501-5. doi: 10.1097/ICO.0000000000000729. PMID 26751993
- [Background] Ozturk Karabulut G, Fazil K. Corneal Topographical Changes After Muller's Muscle-conjunctival Resection Surgery. Ophthalmic Plast Reconstr Surg. 2019 Mar/Apr;35(2):177-181. doi: 10.1097/IOP.0000000000001203. PMID 30130332
- [Background] Zloto O, Matani A, Sagiv O, Prat D, Ben Artsi E, Leshno A, Priel A, Ben Simon GJ. Changes in Refraction and Visual Acuity after Upper Eyelid Blepharoplasty versus Posterior Approach Ptosis Procedures. Ophthalmic Res. 2020;63(6):588-592. doi: 10.1159/000506951. Epub 2020 Mar 5. PMID 32135543
- [Background] Altin Ekin M, Karadeniz Ugurlu S. Prospective analysis of visual function changes in patients with dermatochalasis after upper eyelid blepharoplasty. Eur J Ophthalmol. 2020 Sep;30(5):978-984. doi: 10.1177/1120672119857501. Epub 2019 Jun 17. PMID 31203659
- [Background] Bhattacharjee K, Misra D, Singh M, Deori N. Long-term changes in contrast-sensitivity, corneal topography and higher-order aberrations after upper eyelid blepharoplasty: A prospective interventional study. Indian J Ophthalmol. 2020 Dec;68(12):2906-2910. doi: 10.4103/ijo.IJO_907_20. PMID 33229668
- [Background] Li X, Liu C, Mao Z, Liang X, Li Z, Liu X, Gong R, Huang D. Effect of congenital blepharoptosis on corneal biomechanical properties and changes after ptosis surgery. Eye (Lond). 2020 Jun;34(6):1055-1062. doi: 10.1038/s41433-019-0586-9. Epub 2019 Sep 26. PMID 31558826
- [Background] Sommer F, Untch E, Spoerl E, Herber R, Pillunat LE, Terai N. Effect of upper eyelid blepharoplasty on corneal biomechanical, topographic and tomographic parameters 4 weeks after surgery. Int Ophthalmol. 2022 Jan;42(1):113-121. doi: 10.1007/s10792-021-02006-6. Epub 2021 Sep 3. PMID 34478004
- [Background] Dogan AS, Acar M, Kosker M, Arslan N, Gurdal C. Alterations in corneal epithelial thickness in patients with congenital myogenic eyelid ptosis. Int Ophthalmol. 2018 Feb;38(1):53-57. doi: 10.1007/s10792-016-0419-9. Epub 2016 Dec 26. PMID 28025794
- [Background] Yamamoto R, Ono T, Toyono T, Shirakawa R, Noda M, Yoshida J, Miyai T. Assessment of Long-Term Anterior and Posterior Topographic Changes in the Cornea After Ptosis Surgery Using Fourier Harmonic Analysis. Cornea. 2021 Apr;40(4):440-444. doi: 10.1097/ICO.0000000000002429. PMID 33881809
- [Background] Kanclerz P, Khoramnia R, Wang X. Current Developments in Corneal Topography and Tomography. Diagnostics (Basel). 2021 Aug 13;11(8):1466. doi: 10.3390/diagnostics11081466. PMID 34441401
- [Background] Grubbs JR Jr, Tolleson-Rinehart S, Huynh K, Davis RM. A review of quality of life measures in dry eye questionnaires. Cornea. 2014 Feb;33(2):215-8. doi: 10.1097/ICO.0000000000000038. PMID 24326332
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Ang M, Baskaran M, Werkmeister RM, Chua J, Schmidl D, Aranha Dos Santos V, Garhofer G, Mehta JS, Schmetterer L. Anterior segment optical coherence tomography. Prog Retin Eye Res. 2018 Sep;66:132-156. doi: 10.1016/j.preteyeres.2018.04.002. Epub 2018 Apr 7. PMID 29635068